CLINICAL TRIAL: NCT03447080
Title: Co-ingestion of Rice Bran Soymilk or Plain Soymilk With White Bread: Effects on the Glycaemic and Insulinaemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017/00286
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — soybean-milk-coagulating enzyme

STUDY DESIGN:
Intervention Model Description: Randomized crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control 1 (Other): White bread
  Interventions: Other: Control
- Control 2 (Other): White bread
  Interventions: Other: Control
- Rice bran soybean milk (Experimental): White Bread with 195ml of rice bran soybean mil
  Interventions: Other: Ricebran soybean milk
- Soybean milk (Experimental): White Bread with 195ml of soybean milk
  Interventions: Other: Soybean milk

INTERVENTIONS:
Other: Control — White Bread containing 50g carbohydrate
  Arms: Control 1
Other: Control — White Bread containing 50g carbohydrate
  Arms: Control 2
Other: Ricebran soybean milk — White Bread with rice bran soybean milk
  Arms: Rice bran soybean milk
Other: Soybean milk — White Bread with soybean milk
  Arms: Soybean milk

SUMMARY:
bread and that rice-bran soymilk will have an additional beneficial effect on the glucose and insulin The proposed research project is important because it will provide, for the first time, evidence on the benefits of the addition of rice-bran to soymilk by measuring the acute effect on the glycaemic and insulinaemic response in co-consumption with a high GI meal in Asians. Investigators hypothesize that soymilk will lower the glycaemic and insulinaemic response of white response. This will have an important implication for public health as investigators will understand better how additional dietary fibre can improve the local diet which is typically of high GI values. Ultimately, results from this project will enable the development of dietary recommendations for better glycaemic control in Asian people.

DETAILED DESCRIPTION:
The study will recruit 15-20 young healthy Asian men of Chinese descent. Volunteers will visit Clinical Nutrition Research Centre (CNRC) on 5 occasions: once for consenting and screening procedures (visit 1) and four additional times, interspaced by a minimum of 2 days, to follow a 3 hour test session (Visit 2-5). The study aims to compare the effects of four different test meals , White bread, White bread , Rice-bran soymilk with white bread, Soymilk with white bread, on the glycaemic and insulinaemic response. Visit 1 (screening): For screening, potential subjects will come in the morning after an overnight fast. After obtaining informed consent, a series of screening tests will be conducted, including questionnaires (general health, physical activity and eating behaviour), anthropometry (height, weight, waist and hip circumference), blood pressure, fasting blood glucose, HbA1c and body composition by bioelectrical impedance analysis. Visits 2 to 5 (four experimental trials, in random order): Each of the four study visits will last for approximately 3 hours in the morning, during which the following will take place:During each test session, the subject arrives at the centre between 8:00 and 9:00 in the morning after an overnight fast and has been instructed to avoid any physical activity/exercise and alcohol on the day prior to the test. The session will start by placing an indwelling catheter into a vein in the forearm by trained personnel in a sterile environment. The catheter will be kept patent at all times and left on the forearm until the end of the session. Blood samples will then be taken from the cannula and from a finger prick to measure baseline levels of metabolites. Finger pricks will be done using disposable individual lancets which can cause minimal discomfort. After obtaining baseline blood samples, the subject will be given the test meal to consume within 15 minutes. Following the consumption of the test meal, blood samples (from the cannula and finger pricks) will be collected at periodic intervals (every 15 minutes for the first 90 minutes and every 30 minutes for the remaining 90 minutes). At each time point, a maximum of 5mL of blood will be drawn. In addition, at the same time points, finger prick blood samples will be taken for glucose analysis. At the end of 3 hours of testing, the catheter will be removed and the subject will be free to leave the laboratory. During the entire test session, the subject will have to stay rested and in the laboratory. Television and a workspace will be provided to the subject. In total over the 4 sessions, a maximum of 200 mL of blood (approximately 40 teaspoons) will be collected as part of this study. The blood obtained will be used to measure parameters such as glucose and insulin. Any blood obtained during the course of this study will be stored and analysed for the purposes of this study for a period not exceeding 3 years upon completion of this study. All the study diets will be prepared in the CNRC food preparation kitchen and will use locally sourced ingredients and food purchased from local supermarkets and food distributors.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 21-60 years
* Chinese Ethnicity
* Body mass index between 18.5 - 29 kg/m2
* Fasting blood glucose < 7 mmol/L
* Normal blood pressure (<140/90 mmHg)

Exclusion Criteria:

* have metabolic diseases (such as diabetes, hypertension etc.)
* have glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Currently on prescription medication that may affect metabolism
* Intentionally restrict food intake
* Allergic to wheat bread, rice bran and soya bean

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All healthy male subjects
Enrollment: 17 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Change in postprandial blood glucose over 180 minutes period | 180 minutes
  Blood obtained through fingerprick, analysed using Hemocue analyser.

SECONDARY OUTCOMES:
Change in postprandial plasma insulin over 180 minutes period | 180 minutes
  Venous blood obtain through cannula, analysed using Cobas analyser.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Reseach Centre, Singapore, Singapore